CLINICAL TRIAL: NCT01788683
Title: A Randomized Controlled Trial of Regenexx™ SD Versus Exercise Therapy for Treatment of Non-retracted Supraspinatus Tendon Tears
Brief Title: Regenexx™ SD Versus Exercise Therapy for Rotator Cuff Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regenexx, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RSI2012-RCT01
Record Dates: First submitted 2013-02-06; First posted 2013-02-11 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator Cuff; Rotator Cuff Tear; Supraspinatus Tear
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regenexx SD (Active Comparator): Bone Marrow Aspirate Concentrate injected under imaging guidance into the area of the damaged tendon.
  Interventions: Procedure: Regenexx SD
- Exercise Therapy (Active Comparator): Subjects will be instructed in a set of appropriate rotator cuff strengthening exercises and given an instructional hand-out to take home.
  Interventions: Other: Exercise Therapy

INTERVENTIONS:
Procedure: Regenexx SD — stem cell treatment
  Arms: Regenexx SD
Other: Exercise Therapy — exercise therapy control
  Arms: Exercise Therapy

SUMMARY:
The primary objective of this study is to compare the improvement in subject-reported clinical outcomes, for Regenexx SD treatment vs. Exercise Therapy of non-retracted supraspinatus tendon tears, from baseline to 3 months, with continued evaluation of efficacy and durability up to 24 months.

Secondary objectives include evaluation of US evidence of tendon repair; incidence of post-operative complications, adverse events, re-injections, and surgical intervention; change in pain score and use of pain medications.

DETAILED DESCRIPTION:
Prospective, randomized, controlled to include 34 subjects treated with Regenexx SD and 17 subjects treated with Exercise Therapy alone (2:1 randomization).

Subjects will have a non-retracted supraspinatus tendon tear comprising at least one half the tendon thickness in the anterior-posterior and/or superior-inferior planes as evidenced with positive diagnostic imaging such as arthrogram, ultrasound and/or MR.

Subjects will be enrolled within 60 days prior to Regenexx-SD injection or initiation of exercise therapy and take part in follow-up visits for two years following treatment. A preoperative visit will occur at the time of enrollment; follow-up visits will occur at the clinical site at 6 weeks, 3 months, 6 months, 12 months, and 24 months post injection.

The primary endpoint analysis will be conducted once all subjects reach the 3 month endpoint. At that point, subjects enrolled in the Exercise Therapy group will be given the option of crossing over to the Regenexx SD treatment groups. Subjects will continue to be followed through the 2 year endpoint with data analysis performed at the 1 year and 2 year time points.

Subjects will complete the study following the 2 year follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Physical examination consistent with Rotator Cuff tear
* Unremitting pain in the affected shoulder for at least 3 months
* Significant functional disability related to pain, lack of strength, or other shoulder symptoms
* Positive diagnostic imaging, which may include arthrogram, ultrasound and/or MR, on the affected shoulder indicating a non-retracted supraspinatus tendon tear comprising at least one half the tendon thickness in the anterior-posterior and/or superior-inferior planes
* Reasonable movement of the non-treated arm, defined as a shoulder elevation of equal or more than 90°, and able to perform (post-injection) exercises
* Is independent, ambulatory, and can comply with all post-operative evaluations and visits

Exclusion Criteria:

* A massive rotator cuff tear as demonstrated by Grade 3 or less muscle strength on testing internal and external rotation of the affected shoulder
* Previous surgery to the affected shoulder
* Concomitant tears of biceps tendons
* Grade 2 or greater SLAP tear
* Type 3 acromion
* Significant bone spur in subacromial space
* Inflammatory or auto-immune based joint diseases or other upper extremity pathology (e.g., rheumatoid arthritis, systemic lupus erythematosus, psoriatic arthritis, polymyalgia, polymyositis, gout pseudogout)
* Quinolone or Statin induced myopathy/ tendinopathy
* Kellgren-Lawrence grade 2 or greater glenohumeral osteoarthritis
* Adhesive capsulitis (mild or severe)
* Symptomatic cervical spine pathology (e.g. radicular cervical pain)
* Severe neurogenic inflammation of the cutaneous nerves about the shoulder
* Shoulder instability requiring surgical stabilization
* Contraindications for MRI
* Tested positive or has been treated for a malignancy in the past or is suspected of having a malignancy or is currently undergoing radiation or chemotherapy treatment for a malignancy anywhere in the body, whether adjacent to or distant from the proposed injection site
* Condition represents a worker's compensation case
* Currently involved in a health-related litigation procedure
* Is pregnant
* Bleeding disorders
* Currently taking anticoagulant or immunosuppressive medication
* Use of chronic opioid

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
DASH Score Change from Baseline | Change from Baseline to 3 months
  The primary endpoint for this study is the difference between treatment groups in the within patient mean change from baseline to 3 months in Disabilities of the Arm Shoulder and Hand (DASH) scores.

SECONDARY OUTCOMES:
Mean Pain Scales | 3, 6, 12 and 24 months
  Difference between treatment groups in mean 0-10 pain scales at each follow-up timepoint
MRI evidence of tendon repair | 12 months
  Comparison between groups of MRI evidence of tendon repair at 12 months
Mean DASH scores | 6, 12 and 24 months
  Difference between treatment groups in mean Disabilities of Arm Shoulder and Hand (DASH) scores at 6, 12 and 24 months.
Incidence of Complications and Adverse Events | 24 months
  Incidence and time to resolution of post-operative complications and adverse events between treatment groups.
Incidence of re-injection and surgical revision | 24 months
  Incidence of and time to re-injection and surgical revision between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Centeno, MD, Principal Investigator — Centeno-Schultz Clinic
Locations (1):
- Centeno-Schultz Clinic, Broomfield, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Centeno CJ, Fausel Z, Dodson E, Berger DR, Steinmetz NJ. Percutaneous bone marrow concentrate and platelet products versus exercise therapy for the treatment of rotator cuff tears: a randomized controlled, crossover trial with 2-year follow-up. BMC Musculoskelet Disord. 2024 May 18;25(1):392. doi: 10.1186/s12891-024-07519-6. PMID 38762734
- [Derived] Centeno C, Fausel Z, Stemper I, Azuike U, Dodson E. A Randomized Controlled Trial of the Treatment of Rotator Cuff Tears with Bone Marrow Concentrate and Platelet Products Compared to Exercise Therapy: A Midterm Analysis. Stem Cells Int. 2020 Jan 30;2020:5962354. doi: 10.1155/2020/5962354. eCollection 2020. PMID 32399045